CLINICAL TRIAL: NCT04953247
Title: Use of Compromised Lung Volume in Monitoring Usage of Steroid Therapy on Severe COVID-19
Status: Completed | Type: Observational
Sponsor: Guowei Tu (Other)
Responsible Party: Sponsor-Investigator, Guowei Tu, Scientific Secretary for Department of Critical Care Medcine, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Other Study IDs: CLVMUST
Record Dates: First submitted 2021-07-04; First posted 2021-07-07 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: COVID-19 Pneumonia; Quantitative Computed Tomography
Keywords: Steroid; COVID-19; Quantitative computed tomography; Compromised lung volume
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Methylprednisolone: As there was no consensus on the use of steroids in the early stage of the COVID-19 pandemic, all steroid therapies were initiated at the time of admission at the discretion of attending physicians on the basis of clinical symptoms and CT images. According to our previous experience, intravenous methylprednisolone at a dose of 1.0-1.5 mg/kg every 12 h was initiated for 5 days or until oxygen saturation improved, followed by gradual tapering by 0.5 mg/kg every 3-5 days.
  Standard care such as the use of antibiotics, ventilation, laboratory testing, and hemodynamic management were performed following the sixth edition of the Guidelines on the Diagnosis and Treatment of COVID-19 published by the National Health Commission of China.
- Standard care: Standard care were performed following the sixth edition of the Guidelines on the Diagnosis and Treatment of COVID-19 published by the National Health Commission of China.

SUMMARY:
Since December 2019, the outbreak of coronavirus disease 2019 (COVID-19) has become a public health emergency of international concern. Although corticosteroid therapy represents a milestone in the management of COVID-19, many questions remain unanswered. The optimal type of corticosteroids, timing of initiation, dose, mode of administration, duration, and dose tapering are still unclear. An approach to resolve these issues is to develop accurate tools to assess or monitor the progression of COVID-19 during the corticosteroid therapy process. Quantitative computed tomography (QCT) analysis may serve as a tool for assessing the severity of COVID-19 and for monitoring its progress. However, the effect of steroids on quantitative chest CT parameters during the treatment process remains unknown. In this retrospectively study, we aimed to assess the association between steroid administration and QCT variables in a longitudinal cohort with COVID-19

DETAILED DESCRIPTION:
Since December 2019, the outbreak of coronavirus disease 2019 (COVID-19) has become a public health emergency of international concern. Although corticosteroid therapy represents a milestone in the management of COVID-19, many questions remain unanswered. The optimal type of corticosteroids, timing of initiation, dose, mode of administration, duration, and dose tapering are still unclear. An approach to resolve these issues is to develop accurate tools to assess or monitor the progression of COVID-19 during the corticosteroid therapy process. Quantitative computed tomography (QCT) analysis may serve as a tool for assessing the severity of COVID-19 and for monitoring its progress. However, the effect of steroids on quantitative chest CT parameters during the treatment process remains unknown. In this retrospectively study, we aimed to assess the association between steroid administration and QCT variables in a longitudinal cohort with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* (1) age 18-90 years
* (2) patients with severe or critical COVID-19.

Exclusion Criteria:

* (1) hematological or solid malignancies
* (2) patients with less than two CT scans during hospital stay
* (3) systemic corticosteroid or immunosuppressive therapy in the previous 6 weeks.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From February 7, 2020 to February 17, 2020, consecutive patients with confirmed COVID-19 admitted to the east campus of Renmin Hospital of Wuhan University were screened. The diagnosis of COVID-19 was based on the detection of SARS-CoV-2 nucleic acid by a real-time RT-PCR assay.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Changes in the percentage of compromised lung volume (Δ%CL) at different stages | 31 days
  According to different Hounsfield unit (HU) intervals in the quantitative chest CT scan, we divided each lung into nonaerated lung volume (%NNL, 100 to -100 HU), poorly aerated lung volume (%PAL, -101 to -500 HU), normally aerated lung volume (%NAL, -501 to -900 HU), and hyperinflated lung volume (%HI, -901 to -1000 HU) regions. The additional "compromised lung" volume (%CL) was considered as the sum of %PAL and %NNL (-500 to 100 HU).
  To monitor COVID-19 progression during the treatment process, we chose changes in the percentage of compromised lung volume (Δ%CL) at different stages (Δ%CL = %CL at different stages-baseline %CL) as the primary outcome. The negative value of Δ%CL thus reflected clinical improvement.

SECONDARY OUTCOMES:
Changes in the percentage of NNL at different stages | 31 days
  According to different Hounsfield unit (HU) intervals in the quantitative chest CT scan, we divided each lung into nonaerated lung volume (%NNL, 100 to -100 HU), poorly aerated lung volume (%PAL, -101 to -500 HU), normally aerated lung volume (%NAL, -501 to -900 HU), and hyperinflated lung volume (%HI, -901 to -1000 HU) regions.
Changes in the percentage of PAL at different stages | 31 days
  According to different Hounsfield unit (HU) intervals in the quantitative chest CT scan, we divided each lung into nonaerated lung volume (%NNL, 100 to -100 HU), poorly aerated lung volume (%PAL, -101 to -500 HU), normally aerated lung volume (%NAL, -501 to -900 HU), and hyperinflated lung volume (%HI, -901 to -1000 HU) regions. Under these circumstances, clinical improvement was reflected by the negative value of Δ%NNL and Δ%PAL, and the positive value of Δ%NAL.
Changes in the percentage of NAL at different stages | 31 days
  According to different Hounsfield unit (HU) intervals in the quantitative chest CT scan, we divided each lung into nonaerated lung volume (%NNL, 100 to -100 HU), poorly aerated lung volume (%PAL, -101 to -500 HU), normally aerated lung volume (%NAL, -501 to -900 HU), and hyperinflated lung volume (%HI, -901 to -1000 HU) regions. Under these circumstances, clinical improvement was reflected by the negative value of Δ%NNL and Δ%PAL, and the positive value of Δ%NAL.
Changes in the percentage of HL at different stages | 31 days
  According to different Hounsfield unit (HU) intervals in the quantitative chest CT scan, we divided each lung into nonaerated lung volume (%NNL, 100 to -100 HU), poorly aerated lung volume (%PAL, -101 to -500 HU), normally aerated lung volume (%NAL, -501 to -900 HU), and hyperinflated lung volume (%HI, -901 to -1000 HU) regions. Under these circumstances, clinical improvement was reflected by the negative value of Δ%NNL and Δ%PAL, and the positive value of Δ%NAL.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan hospital, Fudan university, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Su Y, Qiu ZS, Chen J, Ju MJ, Ma GG, He JW, Yu SJ, Liu K, Lure FYM, Tu GW, Zhang YY, Luo Z. Usage of compromised lung volume in monitoring steroid therapy on severe COVID-19. Respir Res. 2022 Apr 29;23(1):105. doi: 10.1186/s12931-022-02025-6. PMID 35488261